CLINICAL TRIAL: NCT01284439
Title: Effect of Hydroxypropylmethylcellulose 0.3% and Sodium Hyaluronate 0.18% in the Treatment of Ocular Surface Disease in Glaucoma Patients
Brief Title: Hydroxypropylmethylcellulose 0.3% and Sodium Hyaluronate 0.18% for Ocular Surface Disease in Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: AssocProf Pinnita Tanthuvanit, Department of Ophthalmology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 655/2553(EC4)
Record Dates: First submitted 2011-01-25; First posted 2011-01-27 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2011-01

CONDITIONS: Ocular Surface Disease; Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Hypromellose Derivatives; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TearA (Experimental)
  Interventions: Drug: hydroxypropylmethylcellulose
- TearB (Experimental)
  Interventions: Drug: sodium hyaluronate

INTERVENTIONS:
Drug: hydroxypropylmethylcellulose — TearA: QID to every 2 hous , 1-2 drops per each time , duration 1 month
  Arms: TearA
Drug: sodium hyaluronate — QID to every 2 hous, 1-2 drops per each time, duration 1 month
  Arms: TearB

SUMMARY:
To study effect of hydroxypropylmethylcellulose 0.3% and sodium hyaluronate 0.18% in the treatment of ocular surface disease in glaucoma patients.

ELIGIBILITY:
Inclusion Criteria:

* OSDI > or equal 20 and eye lid inflammation , meibomian gland inflammation,conjunctival injection,follicle at tarsus , positive corneal staining , tear break up time less than 8 seconds , tear volume less than 5.5 mm.

Exclusion Criteria:

* Age below 18 yo
* Active infectious corneal disease
* Post penetrating keratoplasty or glaucoma drainage device
* Known allergy to medication
* Lactation , Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Ocular surface index score | 1 month

SECONDARY OUTCOMES:
Eye lid inflammation, corneal staining score, tear break up time and tear volume | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: AssocProf Pinnita Tanthuvanit, MD, Principal Investigator — Mahidol University
Locations (1):
- Department of Ophthalmology , Siriraj Hospital, Bangkok, Bangkok, Thailand